CLINICAL TRIAL: NCT07164833
Title: Randomized, Single-blind, Multi-center, Placebo-controlled, Phase 2a Clinical Trial of BX-001N to Prevent From Cardiac Surgery-Associated Acute Kidney Injury (CSA-AKI) and Subsequent Major Adverse Kidney Events (MAKE)
Brief Title: A Study to Evaluate the Efficacy and Safety of BX-001N in Preventing Cardiac Surgery-Associated Acute Kidney Injury (CSA-AKI) and Major Adverse Kidney Events (MAKE)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bilix Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BX-001N-002
Record Dates: First submitted 2025-08-27; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-08

CONDITIONS: Ischemia Reperfusion Injury; Cardiac Surgery Associated - Acute Kidney Injury
MeSH Terms: conditions — Reperfusion Injury

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BX-001N Experimental group 1 (Experimental): Three low doses of BX-001N once a day on the scheduled date
  Interventions: Drug: BX-001N Experimental group 1
- BX-001N Experimental group 2 (Experimental): Three high doses of BX-001N once a day on the scheduled date
  Interventions: Drug: BX-001N Experimental group 2
- Placebo (Placebo Comparator): Three low doses of placebo once a day on the scheduled date
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BX-001N Experimental group 1 — Each participant will receive BX-001N at a weight-based low dose via IV injection once daily for a total of three administrations.
  Arms: BX-001N Experimental group 1
Drug: BX-001N Experimental group 2 — Each participant will receive BX-001N at a weight-based high dose via IV injection once daily at the same time during hospitalization, for a total of three administrations.
  Arms: BX-001N Experimental group 2
Drug: Placebo — Each participant will receive Placebo at a weight-based dose via IV injection once daily at the same time during hospitalization, for a total of three administrations.
  Arms: Placebo

SUMMARY:
This is a Randomized, Single-blind, Multi-center, Placebo-controlled, Phase 2a clinical trial of BX-001N to prevent patients from Cardiac Surgery Associated Acute Kidney Injury (CSA-AKI) and subsequent Major Adverse Kidney Events (MAKE) in approximately 40 participants.

DETAILED DESCRIPTION:
This study will enroll approximately 40 participants, with 16 participants randomized to Experimental Group 1, 16 participants to Experimental Group 2, and 8 participants to the Placebo Group.

Randomized participants will be hospitalized from one day prior to surgery (Baseline, Day -1) through Day 7.

Investigational product (IP) (i.e., BX-001N) will be administered intravenously at a weight-based dose as follows: The test drug will be administered three times in total. Participants in the Placebo Group will receive placebo at the same time points and in the same manner.

Follow-up visits will be conducted up to Day 90 at the study site for scheduled efficacy and safety assessments.

ELIGIBILITY:
Inclusion Criteria:

1. 19 to 90 years of age
2. Participants with aortic disease scheduled for cardiac surgery via total circulatory arrest (TCA)
3. Body weight ≥ 30 kg
4. Participants with vital signs within the following ranges

   * Temperature : 35.0~37.5°C
   * Blood pressure : Systolic blood pressure(SBP) 100~160 mmHg, Diastolic blood pressure(DBP) < 100 mmHg
   * Pulse : 50~100 bpm (regardless of drug use)
5. Willing to comply with the schedule and sign the informed consent

Exclusion Criteria:

1. Participants scheduled for emergent or salvage cardiac surgery
2. Use of kidney replacement therapy (KRT) or presence of acute kidney injury (AKI)
3. Participants with moderate renal impairement
4. Participants at risk of bleeding
5. Participants who underwent cardiac surgery via mid-sternotomy or thoracotomy, including major congenital heart disease
6. Participants who received cardiopulmonary resuscitation within 30 days prior to cardiac surgery
7. Recipient of a solid organ or bone marrow transplantation
8. Participants with cardiogenic shock or hemodynamics instability, or planned use of intra-aortic balloon pump, extracorporeal membrane oxygenation, or left ventricular assist device
9. Active systemic bacterial, viral, or fungal infection
10. History of HIV
11. Positive serology test for HAV, HBV, HCV or Syphilis
12. Participants with impaired liver function due to cirrhosis, or those with 2x UNR blood levels of ALP, AST, or ALT, or with total bilirubin levels outside the normal range
13. Uncontrolled hypertension
14. History of congenital immunodeficiency
15. Genetic disorder with severe and abnormal bilirubin metabolism
16. Participants deemed unsuitable for the study in the discretion of the investigator
17. History of malignancy
18. Planned use of any pharmacologic agent other than the IP assigned in this study for the prevention or treatment of acute kidney injury
19. History of severe allergic or anaphylactic reactions, or sensitivity to the IP or its constituents
20. History of participation in other clinical trials within 30 days
21. Presence of a do-not-resuscitate order or life expectancy of < 3 months
22. Female subjects of childbearing potential
23. Male subjects and their spouse/partner are not willing to use appropriate contraception, or if their spouse/partner is pregnant, breastfeeding or has a plan
24. Poorly controlled type 2 diabetes mellitus
25. New York Heart Association (NYHA) Class IV heart failure

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-26 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in NGAL levels | Baseline(Day -1) to Day 7
Change from baseline in sCr levels | Baseline(Day -1) to Day 7
Change from baseline in eGFR | Baseline(Day -1) to Day 30

SECONDARY OUTCOMES:
Change from baseline in CysC | Baseline(Day -1) to Day 7
Change from baseline in TIMP-2 | Baseline(Day -1) to Day 7
Change from baseline in IGFBP7 | Baseline(Day -1) to Day 7
Collection of Major Adverse Renal Events [MAKE] | Up to Day 90
Change from baseline in Incidence of AKI based on Kidney Disease: Improving Global Outcomes [KDIGO] criteria | Baseline(Day -1) to Day 7
  [Staging of AKI] Stage 1 : 1.5-1.9 times baseline or ≥0.3mg/dL increase Stage 2 : 2.0-2.9 times baseline Stage 3 : 3.0 times baseline or increase in serum creatinine to ≥4.0mg/dL or Initiation of renal replacement therapy
Change from baseline in BUN | Baseline(Day -1) to Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Myung Lip Kim, Chief Executive Officer, Study Chair — Bilix Co.,Ltd.
Locations (5):
- South Korea (5):
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Seoul Asan Medical center, Seoul
  - Pusan National University Yangsan Hospital, Yangsan

IPD SHARING:
Plan to Share IPD: No